CLINICAL TRIAL: NCT04371809
Title: DNA Methylation Analysis to Identify Functional Epigenetic Marks in Acute Coronary Syndrome and Atrial Fibrillation: DIANA Clinical Trial
Brief Title: DNA Methylation Analysis in Acute Coronary Syndrome and Atrial Fibrillation: DIANA Clinical Trial
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Teresa Infante, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: GR-2016-02364785
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Atrial Fibrillation
Keywords: Epigenetics; DNA methylation
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Atrial Fibrillation | interventions — Epigenome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA extracted from CD4+ and CD8+ T cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control subjects
  Interventions: Other: DNA methylome
- subjects with Atrial Fibrillation
  Interventions: Other: DNA methylome
- subjects with Acute Coronary Syndrome
  Interventions: Other: DNA methylome
- subjects with Acute Coronary Syndrome and Atrial Fibrillation
  Interventions: Other: DNA methylome

INTERVENTIONS:
Other: DNA methylome — Epigenomics tools combined with bioinformatic analysis to find and correlate putative useful clinical biomarkers with clinical features

SUMMARY:
Although epigenetics has been identified as one of the most relevant pathophysiological components in the development of cardiovascular diseases, there is still considerable difficulty in finding markers of epigenetic damage useful in clinical practice. Moreover, these markers could be useful to predict the onset and severity of disease as well as to stratify stratification the prognostic risk during the follow-up. The aim of this project will be to evaluate the genome wide DNA methylation status in circulating CD4+ T cells and CD8+ T cells in patients with acute coronary syndromes (ACS), atrial fibrillation (AF) and with ACS in the presence of AF.

DETAILED DESCRIPTION:
Study population will include 20 healthy controls admitted to electrocardiographic control without further cardiological, electrocardiographic and clinical evidence of cardiac pathologies, 20 patients with ACS, and 40 patients with ACS affected or not by AF, recruited at the UTIC of the UOC of Cardiology at the "AORN A. Cardarelli" (Naples, Italy) (Director of the UOC: Dr. Ciro Mauro, as Head of Unit of the study at AORN Cardarelli; assisted by Dr. Antonio Ruocco, Medical Director of Cardiology).

Patients with clinically diagnosed of AF and ACS, in particular unstable angina pectoris (UAP), acute myocardial infarction without ST elevation (NSTEMI) and acute myocardial infarction with ST elevation (STEMI), based on clinical history, symptoms, ECG, biomarkers of damage cardiac, coronary angiography, risk factors and/or other clinical tests according to the guidelines for UAP/ NSTEMI and STEMI, will be recruited at the UTIC of the "AORN A. Cardarelli" (Naples, Italy). All recruited subjects will sign a written informed consent for a blood sampling for non-profit research purposes. Pharmacological therapy, diagnostic information and clinical examination data and medical history will be collected from medical records. Blood samples will be collected during normal clinical practice without taking additional samples from the first day of admission before the use of drugs such as heparin and contrast agents (> 90% of the samples will be collected within a day of acute event). Patients with primary cardiomyopathies, congenital heart disease, valvular diseases, stroke, diabetes mellitus, autoimmune diseases, acute infections, chronic lung infections, COPD, emphysema, pneumoconiosis, asthma, chronic bronchitis, tuberculosis, pleurisy, chronic liver disease and kidney disease, hyperthyroidism or subjects whom will claim an acute febrile illness within 2 weeks, will be excluded from the study.

The collection of whole blood will be carried out from patients and controls during the normal clinical practice. Biological samples will be immediately processed and stored at +4 °C at the regional reference biobank of the U.O.C. of Clinical Immunology and Immunohematology, Transfusion Medicine and Transplantation Immunology with annexed Single Regional Reference Laboratory for Organ Transplant Immunology (LIT) at the Department of Internal Medicine at the University of Campania "Luigi Vanvitelli" (Naples, Italy).

A total of 25 mL of peripheral venous blood will be collected in EDTA tubes and usually processed within 1 hour. Peripheral blood mononuclear cells (PBMNCs) will be isolated by Ficoll gradient using Histopaque®-1077 (Sigma-Aldrich) according to manufacturer's instructions.

CD4+ and CD8+ T lymphocytes will be purified from PBMCs using EasySep™ Human CD4+ T and Cell Isolation Kit and EasySep™ Human CD4+ T Cell Isolation Kit (STEMCELL Technologies), starting by 5x107/mL of PBMNCs, respectively.

Genomic DNA of purified lymphocite subset from each study participant will be isolated immediately after cell isolation using DNeasy Blood & Tissue Kit (Qiagen) according to manufacturer's protocol. DNA concentration and purity will be determined by using NanoDrop spectrophotometer ND-2000 (Thermo Scientific) through the evaluation of the absorbance ratio A260/A280 and DNA integrity checked on 1% agarose gel.

RRB Sequencing and bioinformatic analyses will be performed by an external Service.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinically diagnosed of AF and ACS, in particular unstable angina pectoris (UAP), acute myocardial infarction without ST elevation (NSTEMI) and acute myocardial infarction with ST elevation (STEMI), based on clinical history, symptoms, ECG, biomarkers of damage cardiac, coronary angiography, risk factors and/or other clinical tests according to the guidelines for UAP/ NSTEMI and STEMI

Exclusion Criteria:

Patients with known history of cancer, malignancy disorders, active infections, and chronic or immune-mediated diseases.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include 20 healthy controls admitted to electrocardiographic control without further cardiological, electrocardiographic and clinical evidence of cardiac pathologies, 20 patients with ACS, and 20 patients with ACS and 20 patients with AF and ACS.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
DNA methylation status both of CD4+ and CD8+ cells | 6 months
  DNA methylation profile of patients and controls will be measured both in CD4+ and CD8+ cells collected from peripheral blood by using Reduced Representation Bisulfite Sequencing (RRBS)

SECONDARY OUTCOMES:
Bioinformatics analysis to predict putative novel ACS and AF candidate genes | 3 months
  Bioinformatics analysis will be performed in order to find specific differentially methylated disease genes

OTHER OUTCOMES:
Validation of gene expression | 3 months
  The expression levels of the significant differentially methylated genes will be determined by quantitative real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Infante, Biol.D. Msc., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Cardarelli Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Infante T, Franzese M, Ruocco A, Schiano C, Affinito O, Pane K, Memoli D, Rizzo F, Weisz A, Bontempo P, Grimaldi V, Berrino L, Soricelli A, Mauro C, Napoli C. ABCA1, TCF7, NFATC1, PRKCZ, and PDGFA DNA methylation as potential epigenetic-sensitive targets in acute coronary syndrome via network analysis. Epigenetics. 2022 May;17(5):547-563. doi: 10.1080/15592294.2021.1939481. Epub 2021 Jun 21. PMID 34151742
- [Result] Schiano C, Balbi C, Burrello J, Ruocco A, Infante T, Fiorito C, Panella S, Barile L, Mauro C, Vassalli G, Napoli C. De novo DNA methylation induced by circulating extracellular vesicles from acute coronary syndrome patients. Atherosclerosis. 2022 Aug;354:41-52. doi: 10.1016/j.atherosclerosis.2022.06.1026. Epub 2022 Jul 6. PMID 35830762